CLINICAL TRIAL: NCT06298435
Title: Optimising Ventilatory Strategies by Using Positive Respiratory Integer Measurements
Acronym: OPTIMVSPRIME
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 17536
Record Dates: First submitted 2024-02-12; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Hypoxemia; Hypercapnia; Ventilator Associated Pneumonia; Complication of Anesthesia; Postoperative Complications
MeSH Terms: conditions — Hypoxia; Hypercapnia; Pneumonia, Ventilator-Associated; Postoperative Complications | interventions — Intermittent Positive-Pressure Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GA group: Adult patients having undergone surgery under general anesthesia with IPPV in the UMCG between 01-01-2018 and 01-04-2023
  Interventions: Procedure: Intermittent Positive pressure ventilation

INTERVENTIONS:
Procedure: Intermittent Positive pressure ventilation — Intermittent positive pressure ventilation during general anesthesia for non-cardiac surgery

SUMMARY:
• Background Intermittent Positive Pressure Ventilation is used during general anesthesia but can lead to serious complications. Respiratory parameter settings can be adjusted to minimize the detrimental effects of this unphysiological artificial respiration. Determining optimal ventilator settings is a multifactorial problem with many possible realisations. Knowledge of the relationship of patient outcomes with mathematically identifiable integer sets of ventilator setting parameters may help to understand which effects ventilator settings have on patient outcomes. An exploratory database study can provide a basis for further, prospective, interventional studies to find the optimal combination of ventilator settings.

Main research question

* To determine the relationship between the use of mathematically identifiable integer ventilator parameter sets and patient outcomes
* Design (including population, confounders/outcomes) Retrospective database study of all cases of adult patients undergoing procedures in the UMCG under general anesthesia with IPPV between 01-01-2018 and 01-04-2023. Multivariate and mixed-model analyses, where appropriate, will be corrections for patient specific characteristics such as ASA PS, age, BMI, sex.
* Expected results Using mathematically identifiable integer ventilatory parameter sets improves respiratory and/or hemodynamic patient outcomes.

DETAILED DESCRIPTION:
• Introduction and rationale

Intermittent Positive Pressure Ventilation (IPPV) is required for almost every patient under general anesthesia. It is recognized that IPPV is an unphysiological way of breathing and it can have serious complications when instituted incorrectly. 1 Known complications of IPPV include (but are not limited to) desaturation, atelectasis and baro-/volutrauma.

Many studies have tried to determine the optimal settings for ventilatory parameters during IPPV. 2 Currently, however, it is unknown whether the use of specific ventilatory parameter sets is related to improved outcomes for patients undergoing procedures under general anesthesia.

IPPV is commonly instituted using a set of parameters which determine respiratory characteristics among which are Peak Inspiratory Pressure (PIP), Positive End Expiratory Pressure (PEEP), Plateau Pressure (PlatP) and the Fraction of Inspired Oxygen(FiO2). 3 Adjustment of these parameters allows the clinician to optimize the mechanical characteristics of the artificial respiration of the patient.

IPPV changes intrathoracic pressure in a cyclic way. Pressure increases during inspiration and decreases during expiration. The influence of increased intrathoracic pressure, caused by IPPV, on hemodynamic parameters is well known and is one of the factors used by anesthesiologists when instituting IPPV. IPPV-pressures may both increase or decrease hemodynamic parameters such as cardiac preload and left ventricular wall tension, thus influencing not only oxygenation and decarbonization, but also cardiac output, myocardial oxygen consumption and direct cerebral oxygenation. The relationship between respiration and circulation exhibits complex dynamics and understanding this may help to promote more natural and physiologic breathing patterns, leading to improved oxygenation and reduced respiratory distress.

In addition to direct influence of positive ventilatory pressures on hemodynamic factors the cyclic nature of both IPPV and hemodynamic factors needs to be taken into account when investigating the relationship between IPPV and patient outcomes. When changes in respiratory pressures coincide with related physiological phenomena, each cycle may pose an additive influence on both parameters. Furthermore, coinciding physiological cycles may lead to "respiratory entrainment," where the ventilator-induced breaths becomes asynchronizous with the patient's intrinsic respiratory rhythm, leading to ineffective ventilation and increased risk of lung injury. Additionally, reducing respiratory entrainment may help to reduce the likelihood of mechanical fatigue and stress on the lung tissue, as it avoids repetitive or periodic stress on the respiratory system. Using mathematically identified integer sets as ventilatory parameter settings may reduce the coinciding of respiratory cycles with recurring physiological phenomena. Furthermore, the role of mathematical identification of optimal integer sets for use in ventilator parameters can help find optimal settings to reduce complications from Intermittent Positive Pressure Ventilation

Research question To determine the relationship between the use of mathematically identifiable integer ventilator parameter sets and patient outcomes

METHOD Description study design

This is a retrospective database study. A database search of all cases of adult patients undergoing procedures in the UMCG under general anesthesia with IPPV between 01-01-2018 and 01-04-2023 will be conducted. Researchers will use anonymized data only from the existing patient data records.

This study will investigate the relationship of mathematically identifiable integer sets of ventilator setting parameters during surgery performed under general anesthesia with IPPV. Data will be extracted from the Electronic Patient Database and all data will be handled anonymously.

Parameter integer sets will be identified using probabilistic (or Monte Carlo) algorithms and sieve methods. Non-multifactorial and multifactorial sets will be compared and only non-negative integers will be considered for analysis

Univariate, multivariate regression methods and mixed-model analyses, where appropriate, will be used to determine which integer sets in ventilatory parameter settings during surgery performed under general anesthesia and IPPV are related to patient outcomes such as SpO2 and FiO2/ SpO2-ratio

ELIGIBILITY:
* Inclusion criteria: Adult patients having undergone surgery under general anesthesia with Intermittent Positive Pressure Ventilation in the UMCG between 01-01-2018 and 01-04-2023.
* Exclusion criteria: age <18 years; no use ofIntermittent Positive Pressure Ventilation; not under general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria: Adult patients having undergone surgery under general anesthesia with IPPV in the UMCG between 01-01-2018 and 01-04-2023.
  •
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
SpO2/FiO2 ratio | from start of intermittent positive pressure ventilation until end of intermittent positive pressure ventilation, assessed for a maximum of 24 hours after start of Intermittent Positive Pressure Ventilation
SpO2 | from start of intermittent positive pressure ventilation until end of intermittent positive pressure ventilation, assessed for a maximum of 24 hours after start of Intermittent Positive Pressure Ventilation
etCO2 | from start of intermittent positive pressure ventilation until end of intermittent positive pressure ventilation, assessed for a maximum of 24 hours after start of Intermittent Positive Pressure Ventilation
Blood Pressure | from start of intermittent positive pressure ventilation until end of intermittent positive pressure ventilation, assessed for a maximum of 24 hours after start of Intermittent Positive Pressure Ventilation
Heart Rate | from start of intermittent positive pressure ventilation until end of intermittent positive pressure ventilation, assessed for a maximum of 24 hours after start of Intermittent Positive Pressure Ventilation
Positive end Expiratory Pressure | from start of intermittent positive pressure ventilation until end of intermittent positive pressure ventilation, assessed for a maximum of 24 hours after start of Intermittent Positive Pressure Ventilation
Plateau Pressure | from start of intermittent positive pressure ventilation until end of intermittent positive pressure ventilation, assessed for a maximum of 24 hours after start of Intermittent Positive Pressure Ventilation
Respiration rate | from start of intermittent positive pressure ventilation until end of intermittent positive pressure ventilation, assessed for a maximum of 24 hours after start of Intermittent Positive Pressure Ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Barends, phd, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided